CLINICAL TRIAL: NCT05373966
Title: Delphi Consensus on Robotic Radical Nephroureterectomy Curriculum
Brief Title: Robotic Radical Nephroureterectomy Delphi Consensus
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Hooman Djaladat, Professor of Clinical Urology, University of Southern California
Other Study IDs: UP-22-0032
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Consensus Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delphi Panel: A team of experts in the field of robotic RNU will be invited to participate in the current survey. These experts are identified according to surgical experience, research and academic interest, expertise in running training courses, and participation in live-surgery cases.
  Interventions: Other: Delphi Questionnaire

INTERVENTIONS:
Other: Delphi Questionnaire — An invitation email, including a link to the survey, will be sent to the panel of experts in the field of robotic RNU. The Delphi questionnaire will be administered via Welphi.com.
  In the first survey, panel members will outline the training program for robotic RNU.
  In subsequent surveys, the expert panel will evaluate the modified criteria using a 1 to 5-point Likert scale with space provided for suggested edits and comments. Multiple rounds will be conducted until consensus is reached. After each round of Likert responses, the study team will calculate the agreement and distribution of responses. Likert responses will be dichotomized with positive values indicating agreement and neutral or negative values indicating disagreement.
  For the questions that do not reach a consensus of more than 80% in the first round or need further explanation, additional rounds of the survey may be performed.

SUMMARY:
The aim of this study is to develop a structured training program for robotic radical nephroureterectomy (RNU), based on a Delphi consensus among a panel of experts in this field. A standard questionnaire will be used to obtain experts' opinions on the training steps for robotic RNU.

DETAILED DESCRIPTION:
Upper tract urothelial carcinoma (UTUC) is an uncommon, yet biologically heterogeneous disease that accounts for 5-10% of all urothelial tumors. Radical nephroureterectomy (RNU) with bladder cuff excision is the gold standard for the treatment of UTUC patients. While this procedure is traditionally performed via an open approach, minimally invasive techniques have been used more frequently in recent years. A population-based analysis recently reported an increasing trend in the utilization of robotic RNU from 29% in 2010 to 53% in 2016. Robotic approach not only provides better visualization and optimal exposure during RNU but is also associated with improved perioperative outcomes compared to the open method.

Previous studies have shown that patients treated during the learning phase of a surgeon are at risk of inferior outcomes relative to those treated by experienced surgeons. To overcome such suboptimal outcomes, specific training curriculums have been proposed for some urologic procedures, such as robotic radical prostatectomy, radical cystectomy, and partial nephrectomy. Nevertheless, despite the widespread use of robot for RNU in recent years, no training program is currently available to assist urology residents during their learning process.

This study will provide the first training program for robotic RNU. This curriculum can help to track the progression of the trainee and ensure that defined benchmarks of skills will be reached before the trainee progresses to the next level of difficulty. In addition, it will ultimately improve patients' safety during the learning phase of the urologists.

ELIGIBILITY:
Inclusion Criteria:

* Experts in the field of robotic RNU

Exclusion Criteria:

* Panelists who were not able to commit to all rounds of the modified Delphi process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A team of experts in the field of robotic RNU, who are identified according to surgical experience, research and academic interest, expertise in running training courses, and participation in live-surgery cases.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Degree of consensus | 12 months
  The level of agreement for all statements achieving consensus from the expert panel; consensus is predefined as ≥ 80% of the panel rating a given statement

CONTACTS AND LOCATIONS:
Overall Officials: Hooman Djaladat, MD, Principal Investigator — University of Southern California
Locations (1):
- Hooman Djaladat, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munoz JJ, Ellison LM. Upper tract urothelial neoplasms: incidence and survival during the last 2 decades. J Urol. 2000 Nov;164(5):1523-5. PMID 11025695
- [Background] Roupret M, Babjuk M, Burger M, Capoun O, Cohen D, Comperat EM, Cowan NC, Dominguez-Escrig JL, Gontero P, Hugh Mostafid A, Palou J, Peyronnet B, Seisen T, Soukup V, Sylvester RJ, Rhijn BWGV, Zigeuner R, Shariat SF. European Association of Urology Guidelines on Upper Urinary Tract Urothelial Carcinoma: 2020 Update. Eur Urol. 2021 Jan;79(1):62-79. doi: 10.1016/j.eururo.2020.05.042. Epub 2020 Jun 24. PMID 32593530
- [Background] Kenigsberg AP, Smith W, Meng X, Ghandour R, Rapoport L, Bagrodia A, Lotan Y, Woldu SL, Margulis V. Robotic Nephroureterectomy vs Laparoscopic Nephroureterectomy: Increased Utilization, Rates of Lymphadenectomy, Decreased Morbidity Robotically. J Endourol. 2021 Mar;35(3):312-318. doi: 10.1089/end.2020.0496. Epub 2020 Nov 16. PMID 33081512
- [Background] Lee H, Kim HJ, Lee SE, Hong SK, Byun SS. Comparison of oncological and perioperative outcomes of open, laparoscopic, and robotic nephroureterectomy approaches in patients with non-metastatic upper-tract urothelial carcinoma. PLoS One. 2019 Jan 8;14(1):e0210401. doi: 10.1371/journal.pone.0210401. eCollection 2019. PMID 30620766
- [Background] Thompson JE, Egger S, Bohm M, Haynes AM, Matthews J, Rasiah K, Stricker PD. Superior quality of life and improved surgical margins are achievable with robotic radical prostatectomy after a long learning curve: a prospective single-surgeon study of 1552 consecutive cases. Eur Urol. 2014 Mar;65(3):521-31. doi: 10.1016/j.eururo.2013.10.030. Epub 2013 Oct 31. PMID 24287319
- [Background] Thompson JE, Egger S, Bohm M, Siriwardana AR, Haynes AM, Matthews J, Scheltema MJ, Stricker PD. Superior Biochemical Recurrence and Long-term Quality-of-life Outcomes Are Achievable with Robotic Radical Prostatectomy After a Long Learning Curve-Updated Analysis of a Prospective Single-surgeon Cohort of 2206 Consecutive Cases. Eur Urol. 2018 May;73(5):664-671. doi: 10.1016/j.eururo.2017.11.035. Epub 2017 Dec 19. PMID 29273404
- [Background] Veccia A, Carbonara U, Djaladat H, Mehazin R, Eun DD, Reese AC, Meng X, Uzzo R, Srivastava A, Porter J, Farrow JM, Jamil ML, Rosiello G, Tellini R, Mari A, Al-Qathani A, Rha KH, Wang L, Mastroianni R, Ferro M, De Cobelli O, Hakimi K, Crocerossa F, Ghoreifi A, Cacciamani G, Bhattu AS, Mottrie A, Abdollah F, Minervini A, Wu Z, Simone G, Derweesh I, Gonzalgo ML, Margulis V, Sundaram CP, Autorino R. Robotic vs Laparoscopic Nephroureterectomy for Upper Tract Urothelial Carcinoma: A Multicenter Propensity-Score Matched Pair "tetrafecta" Analysis (ROBUUST Collaborative Group). J Endourol. 2022 Jun;36(6):752-759. doi: 10.1089/end.2021.0587. Epub 2022 Feb 25. PMID 35019760
- [Background] Veccia A, Carbonara U, Derweesh I, Mehrazin R, Porter J, Abdollah F, Mazzone E, Sundaram CP, Gonzalgo M, Mastroianni R, Ghoreifi A, Cacciamani GE, Patel D, Marcus J, Danno A, Steward J, Satish Bhattu A, Asghar A, Reese AC, Wu Z, Uzzo RG, Minervini A, Rha KH, Ferro M, Margulis V, Hampton LJ, Simone G, Eun DD, Djaladat H, Mottrie A, Autorino R. Single-stage Xi(R) robotic radical nephroureterectomy for upper tract urothelial carcinoma: surgical technique and outcomes. Minerva Urol Nephrol. 2022 Apr;74(2):233-241. doi: 10.23736/S2724-6051.21.04247-8. Epub 2021 Mar 29. PMID 33781022
- [Result] Lovegrove C, Novara G, Mottrie A, Guru KA, Brown M, Challacombe B, Popert R, Raza J, Van der Poel H, Peabody J, Dasgupta P, Ahmed K. Structured and Modular Training Pathway for Robot-assisted Radical Prostatectomy (RARP): Validation of the RARP Assessment Score and Learning Curve Assessment. Eur Urol. 2016 Mar;69(3):526-35. doi: 10.1016/j.eururo.2015.10.048. Epub 2015 Nov 14. PMID 26585582
- [Result] Volpe A, Ahmed K, Dasgupta P, Ficarra V, Novara G, van der Poel H, Mottrie A. Pilot Validation Study of the European Association of Urology Robotic Training Curriculum. Eur Urol. 2015 Aug;68(2):292-9. doi: 10.1016/j.eururo.2014.10.025. Epub 2014 Oct 31. PMID 25454612
- [Result] Dell'Oglio P, Turri F, Larcher A, D'Hondt F, Sanchez-Salas R, Bochner B, Palou J, Weston R, Hosseini A, Canda AE, Bjerggaard J, Cacciamani G, Olsen KO, Gill I, Piechaud T, Artibani W, van Leeuwen PJ, Stenzl A, Kelly J, Dasgupta P, Wijburg C, Collins JW, Desai M, van der Poel HG, Montorsi F, Wiklund P, Mottrie A; ERUS Educational Working Group and the YAU Working Group on Robot-assisted Surgery. Definition of a Structured Training Curriculum for Robot-assisted Radical Cystectomy with Intracorporeal Ileal Conduit in Male Patients: A Delphi Consensus Study Led by the ERUS Educational Board. Eur Urol Focus. 2022 Jan;8(1):160-164. doi: 10.1016/j.euf.2020.12.015. Epub 2021 Jan 2. PMID 33402314
- [Result] Larcher A, De Naeyer G, Turri F, Dell'Oglio P, Capitanio U, Collins JW, Wiklund P, Van Der Poel H, Montorsi F, Mottrie A; ERUS Educational Working Group and the Young Academic Urologist Working Group on Robot-assisted Surgery. The ERUS Curriculum for Robot-assisted Partial Nephrectomy: Structure Definition and Pilot Clinical Validation. Eur Urol. 2019 Jun;75(6):1023-1031. doi: 10.1016/j.eururo.2019.02.031. Epub 2019 Apr 9. PMID 30979635